CLINICAL TRIAL: NCT01981837
Title: A Phase 2, Open-Label Trial to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics and Exploratory Clinical Activity of ALN-TTRSC in Patients With Transthyretin (TTR) Cardiac Amyloidosis
Brief Title: Phase 2 Study to Evaluate ALN-TTRSC (Revusiran) in Patients With Transthyretin (TTR) Cardiac Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-TTRSC-002
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2018-03

CONDITIONS: TTR-mediated Amyloidosis
Keywords: RNAi therapeutic
MeSH Terms: interventions — revusiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALN-TTRSC (revusiran) (Experimental)
  Interventions: Drug: ALN-TTRSC (revusiran) for subcutaneous administration

INTERVENTIONS:
Drug: ALN-TTRSC (revusiran) for subcutaneous administration

SUMMARY:
The purpose of this study is to determine the pharmacokinetics, pharmacodynamics and exploratory clinical activity of ALN-TTRSC (revusiran) in Patients with Transthyretin (TTR) Cardiac Amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* TTR cardiac amyloidosis;
* Women of child-bearing potential (WOCBP) must have a negative pregnancy test, cannot be breast feeding, and must be willing to use 2 highly effective methods of contraception;
* Male subjects agree to use appropriate contraception;
* Adequate blood counts, liver, renal and heart function;
* Adequate Karnofsky performance status;
* Adequate New York Heart Association (NYHA) Classification Score;
* Clinically stable on heart medications;
* Adequate 6-minute walk test;
* Willing to give written informed consent and are willing to comply with the study requirements.

Exclusion Criteria:

* Known human immunodeficiency virus (HIV) positive status or known or suspected systemic bacterial, viral, parasitic, or fungal infection;
* Subjects with a history of multiple drug allergies or intolerance to SC injection;
* Received an investigational agent other than tafamidis, diflunisal, doxycycline or tauroursodeoxycholic acid, or an investigational device within 30 days prior to first dose of study;
* Uncontrolled hypertension, ischemic heart disease or cardiac arrhythmia;
* Untreated hypo- or hyperthyroidism;
* Prior major organ transplant;
* Considered unfit for the study by the Principal Investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects experiencing adverse events (AEs), serious adverse events (SAEs) and study drug discontinuation. | Up to 63 days

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ALN-TTRSC (revusiran) (Cmax, tmax, t1/2, AUC, CL, Vss, Vz) | Up to 90 days
Effect of ALN-TTRSC (revusiran) on transthyretin (TTR) (Determination of % Lowering of TTR to pretreatment/Baseline Levels) | Up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jared Gollob, MD, Study Director — Alnylam Pharmaceuticals
Locations (4):
- United States (3):
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Cleveland, Ohio
- Clinical Trial Site, London, United Kingdom